CLINICAL TRIAL: NCT05117970
Title: Artificial Intelligence-assisted Diagnosis and Prognostication in Low Ejection Fraction Using Electrocardiograms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Chin Lin, Assistant Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NDMC2021001
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Left Ventricular Systolic Dysfunction (Disorder)
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to intervention will have access to the screening tool.
  Interventions: Other: AI-enabled ECG-based Screening Tool
- Control (No Intervention): Patients randomized to control will continue routine practice.

INTERVENTIONS:
Other: AI-enabled ECG-based Screening Tool — Primary care clinicians in the intervention group had access to the report, which displayed whether the AI-ECG result was positive or negative.The system will send a message to corresponding physicians if positive finding.
  Arms: Intervention

SUMMARY:
This is a randomized controlled trial (RCT) to test a novel artificial intelligence (AI)-enabled electrocardiogram (ECG)-based screening tool for improving the diagnosis and management of left ventricular systolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with EF>50% or without Transesophageal Echocardiography (TEE)

Exclusion Criteria:

* Patients with a history of heart failure or an EF<= 35%.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13631 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
New Diagnosis of Low Ejection Fraction(defined as ejection fraction ≤50%) | Within 30 days
  Ejection fraction obtained by echocardiography

SECONDARY OUTCOMES:
All cause mortality(death) | Within 30 days
  After performing an electrocardiogram, the patient's survival is tracked.
Completion of an echocardiogram | Within 30 days
  After performing the ECG examination, perform the echocardiogram examination

CONTACTS AND LOCATIONS:
Locations (1):
- National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsai DJ, Lin C, Liu WT, Lee CC, Chang CH, Lin WY, Liu YL, Chang DW, Hsieh PH, Tsai CS, Chen YH, Hung YJ, Lin CS. Artificial intelligence-assisted diagnosis and prognostication in low ejection fraction using electrocardiograms in inpatient department: a pragmatic randomized controlled trial. BMC Med. 2025 Jun 9;23(1):342. doi: 10.1186/s12916-025-04190-z. PMID 40484925